CLINICAL TRIAL: NCT04326413
Title: Artificial Intelligence Evaluation of Periodontal Health Using Selfie Intraoral Photography
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Walter Y.H. Lam, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: HKWC-2019-0666
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Oral hygiene instruction and simple scaling — Monitor the changes of gum condition

SUMMARY:
Periodontal (gum) disease affecting more than 90% of the population globally. The soft and hard tissues that supporting the teeth are being affected. If untreated, the disease progresses from the mild and reversible form (i.e. gingivitis) that involves superficial gum only to the more severe and irreversible form (i.e. periodontitis) that involves loss of periodontal ligament and bone. Teeth will be lost eventually and significantly impairs the function and the oral health related quality of health. Moreover, periodontal disease has been strongly linked to the systemic diseases via centrally or local routes with significant health implications.

Periodontal disease is initiated by bacteria (plaque) adhere on tooth surfaces and the body defense by eliciting inflammatory response. The disease and associated inflammation is site-specific and the affected gum is manifested with the cardinal signs of inflammation such as redness (color), swelling (increased volume), edema (loss of surface characteristics) and bleeds easily. Dentists are trained to identify the disease sites by visual (redness and swelling) and by mechanical probing (bleeding). Traditionally these give rises to clinical gum indices showing the degree of inflammation and are important to the clinical monitoring and management of gum diseases.

The management of periodontal disease involves the removal of bacteria plaque by both dentists' tooth cleaning and maintained by patients' daily home-care. Home-care plaque removal has been shown by many studies to prevent and/or cease the development of periodontitis. However, most patients do not able to remove plaque effectively and it only takes few days for a health site to development inflammation. Professional monitoring and feedback are highly desirable but many patients only have monthly or even yearly appointment which is too late. Such "non-compliance" increase the treatment cost/time, patient discomfort and reduce treatment efficacy. Moreover, many patients do not receive regular dental checkup and they seek dentists when the gum problem becomes irreversible that complicated and expensive treatment such as tooth extraction and rehabilitation is required.

This study consists of 1) collecting the standardized clinical photography with clinical gum indices/ marked by an experienced clinician, 2) import into computer for training, and 3) longitudinally monitoring and analyze of gum condition in a group of gingivitis patients receiving gum treatment.

DETAILED DESCRIPTION:
The first part of this study will collect buccal view of intraoral photo and clinical gum indices from 300 patients visiting Prince Philip Dental Hospital (PPDH). These intraoral photo will be taken by patients using smartphone (iphone) mounted with apparatus (Scanbox) in a standardized way and the quality supervised by clinical staff. Clinical gum indices will be taken by a trained and calibrated clinical staff. Alternatively clinical photo may be assessed by an experienced clinician to locate the inflamed/health gum. This synthesized data set imported into neural network to learn the image characteristics of inflamed and health gum and train the computer.

The second part of this study will recruit 150 patients with gingivitis and longitudinally follow up their gum condition pre- and post- gum treatment in PPDH using standardized intraoral photo and clinical gum indices. The clinical gum indices are the gold standard reflecting the changes in the gum condition.

All photos collected would be analyzed by computer (software: MatLab) to identify key features that help with screening and monitoring of gum condition. Data would then be collected for building a program that quantifies the identified features which may include the following:

1. Color of marginal gum tissues
2. Texture of marginal gum tissues
3. Volume of marginal gum tissues, with reference to the clinical gum indices.

Data and sample size analysis: The computer will be trained with the photo and clinical indices/assessment obtained in the part I of this study. The trained computer will then use to monitor changes of periodontal condition of patients in part II of this study based on photo only. The sensitivity (detect true disease), specificity (detect true health) and the area under these curves (with reference to the gold standard clinical gum indices) will be calculated and are the main outcome of this study. The training of computer is a continuous process and the endpoint comes when the sensitivity, specificity and the area under these curves (AUC) reach plateau (saturation). Therefore, the training of computer will be staged into three phrases with 100, 200 and 300 of cases in the part I of this study and observe the changes in the sensitivity, specificity and AUC.

Patient reported outcome on the use of smartphone selfie would be recorded in visual analogue scale (VAS) as secondary outcome.

Sample size determination: Each tooth represents one unit and assume each subject has 20 teeth, there will be more than 300 subjects X 20 teeth =6000 units for training. For the part 2 study, 150 subjects will be recruited and 130X20=2600 units for testing of the computer.

All new patients attending Prince Philip Dental Hospital will be screen for gum inflammation and periodontal diseases by clinical examination.

Basic periodontal examination (BPE, including visual examination and mechanical probing of gum) will be performed for all of them and assign to the undergraduate students for patient care according to the severity.

Computer record can retrieve patients with gum inflammation (BPE score 2). Data handling All data will be kept reviewed by unblended member (YHL) to check the quality. Only the data that related to the study outcomes will be disclosed. All the data will be kept for another two years since the study finishes. After that, the data will be destroyed completely. Primary investigator will have access to the personal data during and after the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects attending PPDH and are able to give informed consent
* Subjects who diagnosed to have gingivitis only and have 24 or more teeth
* Subjects who are otherwise medically health
* Subjects who are able to attend multiple dental visits

Exclusion Criteria:

* Subjects who are in acute dental infection or in pain
* Subjects who have oral mucosal diseases that preclude retraction of soft tissues for photos
* Subjects who are in fixed appliance for orthodontic treatment
* Subjects who are pregnancy, or medically unfit for periodontal charting or requires antibiotic coverage (e.g. risk of infective endocarditis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy dentate patients with gingivitis only and have 24 or more teeth
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Clinical gingival inflammation at 3 month | 3-month
  Mean number/Percentage of sites with, as determined by the plaque index (Silness and Loe 1965 from 0 to 3) by observation of patient's mouth
Photographic gingival inflammation at 3 month | 3-month
  Mean number/Percentage of sites with, as determined by the plaque index (Silness and Loe 1965 from 0 to 3) by observation of patient's standardized photo
Photographic gingival inflammation at baseline | baseline
  Mean number/Percentage of sites with, as determined by the plaque index (Silness and Loe 1965 from 0 to 3) by observation of patient's standardized photo
Clinical gingival inflammation at baseline | baseline
  Mean number/Percentage of sites with, as determined by the plaque index (Silness and Loe 1965 from 0 to 3) by observation of patient's mouth

SECONDARY OUTCOMES:
Patient reported outcome on the use of smartphone selfie | 3-month
  Satisfactory in Visual analogue scale (VAS) from 0 (not satisfactory) to 100 (satisfactory)

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Philip Dental Hospital, Sai Ying Pun, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided